CLINICAL TRIAL: NCT00002766
Title: A Phase III Trial Comparing ARA-C/High-Dose Mitoxantrone ("ALL-2') to A Standard Vincristine/Prednisone Based Regimen ('L-20') as Induction Therapy For Adult Patients With Acute Lymphoblastic Leukemia (ALL): The ALL-4 Protocol
Brief Title: Comparison of Two Combination Chemotherapy Regimens in Treating Adults With Previously Untreated Leukemia or Lymphoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 96-015; P30CA008748 (NIH); MSKCC-96015A1; NCI-V96-0881
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Results first posted 2016-02-22 (Estimated); Last update posted 2016-02-22 (Estimated); Status verified 2016-01

CONDITIONS: Leukemia; Lymphoma
Keywords: blastic phase chronic myelogenous leukemia; untreated adult acute lymphoblastic leukemia; chronic myelogenous leukemia, BCR-ABL1 positive; T-cell adult acute lymphoblastic leukemia; B-cell adult acute lymphoblastic leukemia; stage I adult lymphoblastic lymphoma; stage II adult lymphoblastic lymphoma; stage III adult lymphoblastic lymphoma; stage IV adult lymphoblastic lymphoma; contiguous stage II adult lymphoblastic lymphoma; noncontiguous stage II adult lymphoblastic lymphoma
MeSH Terms: conditions — Leukemia; Lymphoma; Blast Crisis; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Dactinomycin; sargramostim; Carmustine; Cyclophosphamide; Cytarabine; Daunorubicin; Doxorubicin; Etoposide; Mercaptopurine; Methotrexate; Mitoxantrone; pegaspargase; Prednisone; Vincristine; Radiotherapy

ARMS (2):
- ARA-C/High-Dose Mitoxantrone("All-2") (Experimental): See detail description
  Interventions: Biological: dactinomycin; Biological: sargramostim; Drug: carmustine; Drug: cyclophosphamide; Drug: cytarabine; Drug: doxorubicin hydrochloride; Drug: etoposide; Drug: mercaptopurine; Drug: methotrexate; Drug: mitoxantrone hydrochloride; Drug: pegaspargase; Drug: prednisone; Drug: vincristine sulfate; Radiation: radiation therapy
- Standard Vincristine/Prednisone ("L-20") (Active Comparator): See detail description
  Interventions: Biological: sargramostim; Drug: carmustine; Drug: cyclophosphamide; Drug: cytarabine; Drug: daunorubicin hydrochloride; Drug: doxorubicin hydrochloride; Drug: methotrexate; Drug: pegaspargase; Drug: prednisone; Drug: vincristine sulfate

INTERVENTIONS:
Biological: dactinomycin
  Arms: ARA-C/High-Dose Mitoxantrone("All-2")
Biological: sargramostim
Drug: carmustine
Drug: cyclophosphamide
Drug: cytarabine
Drug: daunorubicin hydrochloride
  Arms: Standard Vincristine/Prednisone ("L-20")
Drug: doxorubicin hydrochloride
Drug: etoposide
  Arms: ARA-C/High-Dose Mitoxantrone("All-2")
Drug: mercaptopurine
  Arms: ARA-C/High-Dose Mitoxantrone("All-2")
Drug: methotrexate
Drug: mitoxantrone hydrochloride
  Arms: ARA-C/High-Dose Mitoxantrone("All-2")
Drug: pegaspargase
Drug: prednisone
Drug: vincristine sulfate
Radiation: radiation therapy
  Arms: ARA-C/High-Dose Mitoxantrone("All-2")

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells. It is not yet known which regimen of combination chemotherapy is more effective for acute lymphoblastic leukemia, lymphoblastic lymphoma, or chronic myelogenous leukemia.

PURPOSE: This randomized phase III trial is studying two different chemotherapy regimens and comparing them to see how well they work in treating adults with acute lymphoblastic leukemia, lymphoblastic lymphoma, or chronic myelogenous leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the incidence of complete remission (CR) following induction with the ALL-2 regimen (cytarabine and high-dose mitoxantrone) vs the L-20 regimen (vincristine and prednisone) in previously untreated adult patients with acute lymphoblastic leukemia (ALL), lymphoblastic lymphoma, and lymphoid blast crisis chronic myelogenous leukemia.
* Compare the time to CR, length of hospital stay, efficacy of treatment in Philadelphia chromosome-positive ALL, and the proportion of patients achieving durable (greater than 5 years) remission in each treatment regimen.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to participating institution and antecedent lymphoid blast crisis of chronic myelogenous leukemia (yes vs no). Patients are randomized to one of two treatment arms.

Arm I:

* Patients receive induction therapy consisting of cytarabine IV over 3 hours on days 1-5 with high-dose mitoxantrone IV on day 3 and methotrexate intrathecally on days 2 and 4. Patients receive sargramostim (GM-CSF) subcutaneously or IV over 4 hours beginning on day 7 and continuing until blood counts recover.
* At 7-14 days following induction therapy, patients receive consolidation therapy consisting of vincristine IV on days 1, 8, 15, 22, and 29, oral prednisone 2-3 times daily on days 1-30 and methotrexate intrathecally on days 8, 15, 22, and 29.
* At 2-3 weeks following the last dose of vincristine, patients receive an additional course of consolidation therapy consisting of cyclophosphamide IV on day 1 and GM-CSF subcutaneously beginning on day 3 and continuing until blood counts recover.
* At 3-4 weeks following the second consolidation course, patients receive a third course of consolidation therapy consisting of cytarabine IV bolus on day 1 followed by continuous infusion cytarabine on days 1-4 with etoposide IV over 1 hour on days 1-3 and methotrexate intrathecally on days 2 and 4. Patients receive GM-CSF subcutaneously beginning on day 6 and continuing until blood counts recover.
* Following recovery from the third consolidation course, patients receive a fourth consolidation course consisting of pegaspargase IV or intramuscularly (IM) on day 1.
* Following recovery from consolidation therapy patients receive 2 sequences of maintenance therapy with sequence one consisting of vincristine IV on days 1 and 8, oral prednisone 2-3 times daily on days 1-8, doxorubicin IV on day 15, oral mercaptopurine 2-3 times daily on days 36-64, oral methotrexate on days 39, 46, 53, and 60, dactinomycin IV on day 85, and methotrexate intrathecally on days 36 and 43.
* At 2 weeks following sequence one of maintenance therapy, patients receive sequence two consisting of the same regimen as in the first sequence with the addition of cyclophosphamide IV and carmustine IV on day 15.
* Patients with CNS involvement receive whole brain radiotherapy in addition to chemotherapy regimens.

Arm II:

* Patients receive induction therapy consisting of vincristine IV on days 1, 8, 15, 22, and 29, oral prednisone 2-3 times daily on days 1-29, cyclophosphamide IV on day 5, doxorubicin IV on days 23-25 and 42, methotrexate intrathecally on days 3, 5, 13, 16, 32, and 34 and GM-CSF subcutaneously or IV over 4 hours beginning from days 7 and 27 and continuing until blood counts recover.
* At approximately 3 weeks following induction therapy, patients receive consolidation therapy consisting of cytarabine IV bolus on day 1 followed by continuous infusion cytarabine on days 1-5, with daunorubicin IV on days 1-3 and methotrexate intrathecally on days 2 and 4. Patients receive GM-CSF subcutaneously beginning on day 7 and continuing until blood counts recover.
* At 6-8 weeks following the first course of consolidation therapy, patients receive a second consolidation course consisting of cytarabine IV bolus on day 1 followed by continuous infusion cytarabine on days 1-4 with methotrexate IV on days 1-4 and methotrexate intrathecally on days 2 and 4. Patients receive GM-CSF subcutaneously beginning on day 6 and continuing until blood counts recover.
* At 6-8 weeks following the second course of consolidation therapy, patients receive a third consolidation course consisting of pegaspargase IV or IM on day 1.
* At 3-4 weeks following the third course of consolidation therapy, patients receive a fourth consolidation course consisting of cyclophosphamide IV on day 1.
* At 3 weeks following the completion of consolidation therapy, patients receive the same maintenance regimen as in Arm I.

Treatment continues in patients achieving complete response. Patients in both arms receive alternating sequences of maintenance therapy over 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of one of the following malignancies:

  * Acute lymphoblastic leukemia (ALL) of B- or T-cell lineage
  * Philadelphia chromosome-positive ALL eligible
  * Lymphoblastic lymphoma
  * Chronic myelogenous leukemia in lymphoid blast crisis

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 20-100%

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Bilirubin no greater than 2.0 mg/dL
* Glucocorticoids for higher bilirubin allowed prior to entry, at principal investigator's discretion

Renal:

* Creatinine no greater than 2.0 mg/dL
* Glucocorticoids or renal radiotherapy for higher creatinine allowed prior to entry, at principal investigator's discretion

Cardiovascular:

* Left ventricular ejection fraction at least 50%

Other:

* Not pregnant

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No prior biologic therapy

Chemotherapy

* No prior chemotherapy

Endocrine therapy

* No prior endocrine therapy

Radiotherapy

* No prior radiotherapy

Surgery

* No prior surgery

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 1996-03; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Lamanna, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Stanford Cancer Center at Stanford University Medical Center, Stanford, California
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - New York Medical College, Valhalla, New York
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio

RESULTS

PARTICIPANT FLOW:
Groups:
- All-2: ARA-C/High-Dose Mitoxantrone("All-2") Patients receive induction therapy consisting of cytarabine IV over 3 hours on days 1-5 with high-dose mitoxantrone IV on day 3 and methotrexate intrathecally on days 2 and 4. Patients receive sargramostim (GM-CSF) subcutaneously or IV over 4 hours beginning on day 7 and continuing until blood counts recover.
- L-20: Standard Vincristine/Prednisone ("L-20") Patients receive induction therapy consisting of vincristine IV on days 1, 8, 15, 22, and 29, oral prednisone 2-3 times daily on days 1-29, cyclophosphamide IV on day 5, doxorubicin IV on days 23-25 and 42, methotrexate intrathecally on days 3, 5, 13, 16, 32, and 34 and GM-CSF subcutaneously or IV over 4 hours beginning from days 7 and 27 and continuing until blood counts recover.
Period: Overall Study
Arm/Group | All-2 | L-20
Started | 81 | 89
Completed | 78 | 85
Not Completed | 3 | 4
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Patient Not Treated | 1 | 2
Not completed — Adverse Event | 1 | 1
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- All-2: ARA-C/High-Dose Mitoxantrone("All-2")
- L-20: Standard Vincristine/Prednisone ("L-20")
- Total: Total of all reporting groups
Arm/Group | All-2 | L-20 | Total
Number analyzed (Participants) | 81 | 89 | 170
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3 | 4 | 7
  Between 18 and 65 years | 76 | 77 | 153
  >=65 years | 2 | 8 | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 36 | 67
  Male | 50 | 53 | 103

OUTCOME MEASURES:

1. Primary Outcome: Complete Remission (CR)
Description: complete remission (CR) Disappearance of all clinical evidence of leukemia for a minimum of four weeks. The patient should have a neutrophil count > 1,000 x 10^6/1, a platelet count > 100,000 x 10^9/1, no circulating blasts, and < than or = to blasts on bone marrow differential in a qualitatively normal or hypercellular marrow. Progressive disease or failure: Increasing bone marrow infiltrate or development of organ failure or extramedullary infiltrates due to leukemia.
Time Frame: 2 years
Measure: Number; unit: participants
Arm/Group | All-2 | L-20
Number analyzed (Participants) | 78 | 85
participants
  Complete Remission | 50 | 50
  Complete Response (CR) | 14 | 11
  Failure | 5 | 14
  Failure-Progression | 8 | 10
  Relapse | 1 | 0

ADVERSE EVENTS:
Arm/Group | All-2 | L-20
Serious Adverse Events (participants affected / at risk) | 39/81 | 33/89
Other Adverse Events (participants affected / at risk) | 49/81 | 42/89
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All-2 (N=81) | L-20 (N=89)
Adult respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2)
Abdominal pain/cramping (Gastrointestinal disorders) | 3 (3) | 0 (0)
Acidosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Amylase (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Ataxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Bilirubin (Metabolism and nutrition disorders) | 3 (4) | 1 (1)
Blood,Bone marrow,other (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Bone pain (General disorders) | 1 (1) | 0 (0)
Cardiac left ventricle (Cardiac disorders) | 1 (1) | 0 (0)
Cardiovascular, other (Cardiac disorders) | 1 (1) | 0 (0)
Colitits (Gastrointestinal disorders) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 3 (3) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Dysphagia, esophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Febrile neutropenia (General disorders) | 11 (13) | 13 (17)
Fever (General disorders) | 2 (2) | 0 (0)
Fibrinogen (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hand-Foot Skin reaction (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Headache (General disorders) | 1 (1) | 1 (1)
Hematuria (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hemoglobin (Hgb) (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Hemorrhage, other (General disorders) | 1 (1) | 3 (3)
Hepatic enlargement (Renal and urinary disorders) | 1 (1) | 0 (0)
Hepatic, other (Renal and urinary disorders) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypotension (Cardiac disorders) | 2 (2) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Ileus (or neuroconstipation) (Gastrointestinal disorders) | 1 (1) | 5 (5)
infection (Infections and infestations) | 1 (1) | 2 (2)
Infection with grade 3/4 neutrophils (Infections and infestations) | 1 (1) | 0 (0)
Infection/Febrible Neutrophil-Other (Infections and infestations) | 10 (12) | 4 (4)
Leukocytes (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Neurology, other (Nervous system disorders) | 2 (2) | 0 (0)
Neuropathy-motor (Nervous system disorders) | 2 (2) | 2 (2)
Neutrophils (Leukemia) (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Pain, other (General disorders) | 1 (1) | 2 (2)
Pancreatitis (Gastrointestinal disorders) | 3 (3) | 1 (1)
Platelets (Blood and lymphatic system disorders) | 3 (4) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary, other (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Renal failure (Renal and urinary disorders) | 4 (4) | 2 (2)
SGOT (AST) (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
SGPT (ALT) (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Syncope (General disorders) | 2 (2) | 1 (1)
Ventricular arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Vision-blurred vision (Eye disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Supravent arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Stomatitis/pharyngitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Neutrophils (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Gastrointestinal, other (Gastrointestinal disorders) | 0 (0) | 1 (1)
Epistaxis (General disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2)
Dermatology, skin other (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dehydration (General disorders) | 0 (0) | 2 (2)
disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 1 (1)
Cardiovascular, Arrhythmia other (Cardiac disorders) | 0 (0) | 1 (1)
Ascites (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
ALT, SGPT (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All-2 (N=81) | L-20 (N=89)
Abdominal pain/cramping (Gastrointestinal disorders) | 11 (11) | 12 (12)
Anorexia (General disorders) | 6 (6) | 5 (5)
Bilirubin (Metabolism and nutrition disorders) | 9 (9) | 6 (6)
Bone pain (General disorders) | 6 (6) | 0 (0)
Dizziness (Nervous system disorders) | 7 (7) | 6 (6)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 7 (7)
Fatigue (General disorders) | 12 (12) | 15 (15)
Febrile neutropenia (General disorders) | 7 (7) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 18 (18) | 14 (14)
Hypomagnesemia (Metabolism and nutrition disorders) | 10 (10) | 7 (7)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 5 (5)
Hypophosphatemia (Metabolism and nutrition disorders) | 12 (12) | 13 (13)
Insomnia (General disorders) | 5 (5) | 0 (0)
Muscle weakness (General disorders) | 6 (6) | 0 (0)
Pain, other (General disorders) | 12 (12) | 12 (12)
Prothrombin Time (Blood and lymphatic system disorders) | 0 (0) | 5 (5)
Rigors, chills (General disorders) | 7 (7) | 0 (0)
SGPT (ALT) (Blood and lymphatic system disorders) | 6 (6) | 5 (5)
Stomatitis/pharyngitis (Gastrointestinal disorders) | 5 (5) | 10 (10)
Syncope (Nervous system disorders) | 6 (6) | 0 (0)
Thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 7 (7)
Vision-blurred vision (Eye disorders) | 0 (0) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes